CLINICAL TRIAL: NCT01834924
Title: Dissemination of a Health Literacy Intervention to Improve Provider-Patient Communication of Medication Instructions and Decrease Outpatient Pediatric Medication Errors
Brief Title: Improving Communication of Medication Instructions to Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: New York City Health and Hospitals Corporation (Other); Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: 08-1423
Record Dates: First submitted 2013-04-15; First posted 2013-04-18 (Estimated); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Medication Errors; Medication Adherence
Keywords: Health literacy; Patient education
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HELPix (Active Comparator): Low literacy, bilingual (English/Spanish) medication instruction sheets used as a framework for provider medication counseling, plus provider dose demonstration, parent teachback/showback, provider medication log review, provision of oral dosing syringe to parent
  Interventions: Other: HELPix
- Control (No Intervention): Standard provider medication counseling

INTERVENTIONS:
Other: HELPix — Low literacy, bilingual (English/Spanish) medication instruction sheets used as a framework for provider medication counseling, plus provider dose demonstration, parent teachback/showback, provider medication log review, provision of oral dosing syringe to parent
  Arms: HELPix

SUMMARY:
Almost half of all US adults have trouble understanding and using health information, or low health literacy. Health literacy is considered to be an important patient safety issue, and has been linked to poor medication management. Low health literacy is a risk factor for parent errors in administering medications to their children; difficulty understanding provider medication instructions is likely to contribute to errors.

To address these issues, bilingual (English/Spanish), low literacy, picture-based medication instruction sheets were developed. This study will look at the effectiveness and feasibility of the medication instruction sheet-based intervention as it is used by providers in 2 pediatric emergency department settings, as part of a planned roll out of HELPix within the hospital system. The investigators hypothesize that there will be reduced medication dosing errors, improved medication adherence, reduced hospital revisit rates, and improved provider-parent communication. The investigators also hypothesize that provider technology experience, knowledge, and attitudes, will affect the extent to which providers use the tool.

ELIGIBILITY:
Parent Inclusion Criteria:

* child <=8 years
* child prescribed a daily dose short course (<14 day) liquid medication

Parent Exclusion Criteria:

* caregiver not legal guardian of child
* caregiver non-English/ Spanish language
* caregiver residency outside of New York City
* hospital admission of child
* child with psychiatric or child protection-related issue
* no listed phone number for caregiver
* person reached by phone not person counseled in the emergency department
* no eligible medication prescribed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1196 (Actual)
Dates: Start 2010-05-31 (Actual); Primary Completion 2015-01-09 (Actual); Study Completion 2015-01-09 (Actual)

PRIMARY OUTCOMES:
Medication dosing error (observed) | within 8 weeks of the end date of prescribed course of medication
  Dosing error defined as >20% deviation from prescribed dose

CONTACTS AND LOCATIONS:
Overall Officials: H. Shonna Yin, MD, MS, Principal Investigator — NYU School of Medicine / Bellevue Hospital Center
Locations (2):
- United States (2):
  - Woodhull Hospital, Brooklyn, New York
  - Bellevue Hospital Center, New York, New York